CLINICAL TRIAL: NCT02068469
Title: Multi-Center Study of an In Vitro Diagnostic Device for the Detection of Strep A
Brief Title: In Vitro Diagnostic Device for the Detection of Strep A
Status: Completed | Type: Observational
Sponsor: IQuum, Inc. (Industry)
Collaborators: Roche Molecular Systems, Inc (Industry)
Responsible Party: Sponsor
Other Study IDs: SASA 4.0
Record Dates: First submitted 2014-02-14; First posted 2014-02-21 (Estimated); Last update posted 2016-08-31 (Estimated); Status verified 2016-08

CONDITIONS: Streptococcal Sore Throat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Throat culture swab
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this trial is to show the accuracy and specificity of the Liat analyzer and assay for detecting Strep A at the point of care lab compared to culture.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are 3 years of age or older
* Subjects exhibiting symptoms characteristic of pharyngitis, possibly Streptococcus A, including:

  * presence of sore throat, and at least one other symptom from the list below:
  * redness of the posterior pharyngeal wall
  * pharyngeal or tonsillar exudate
  * tonsillar swelling
  * tender cervical lymphadenopathy
  * fever, >38C at presentation or within the past 24 hours
* Subjects who are able to understand and consent to participation; for minors under the age of 18, this includes parent or legal guardian

Exclusion Criteria:

* Subjects treated with antibiotics currently or within the previous 7 days.

Min Age: 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and Pediatric primary care clinic, walk in clinic
Sampling Method: Non-Probability Sample
Enrollment: 799 (Actual)
Dates: Start 2013-12; Primary Completion 2014-04 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
Evaluate sensitivity and specificity of the Liat Strep A assay when compared to culture | Results based on samples collected at initial visit

CONTACTS AND LOCATIONS:
Overall Officials: Lingjun Chen, BS, Study Director — IQuum COO
Locations (5):
- United States (5):
  - Norwich Pediatrics, Norwich, Connecticut
  - Meridian Clinical Research, Savannah, Georgia
  - Twelve Corners Pediatrics, Rochester, New York
  - Plano Pediatrics, Plano, Texas
  - Advanced Pediatrics, Vienna, Virginia

IPD SHARING:
Plan to Share IPD: No